CLINICAL TRIAL: NCT05618327
Title: Phase I Clinical Study of JS203 in Patients With Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS203-001-I
Record Dates: First submitted 2022-10-20; First posted 2022-11-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS203 (Experimental)
  Interventions: Drug: JS203 for Injection

INTERVENTIONS:
Drug: JS203 for Injection — 2-steps:JS203 for Injection is administered on the first and eighth day of the first cycle and every 3 weeks thereafter.
  3-steps:JS203 for Injection is administered on the first, eighth and fifteenth day of the first cycle and every 3 weeks thereafter.
  4-steps:JS203 for Injection is administered on the first, eighth, fifteenth and twenty-second day of the first cycle and every 3 weeks thereafter.

SUMMARY:
This is an open phase I clinical study to evaluate the safety, tolerability, pharmacokinetic (PK) profile, pharmacodynamic (PD) profile, immunogenicity, and preliminary efficacy of JS203 in patients with relapsed/refractory B-cell non-Hodgkin's lymphoma. The study is divided into three phases: a dose-escalation phase, a dose-expansion phase, and an efficacy expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form.
2. Age 18 - 75 years (both 18 and 75 years), both sexes
3. Expected survival of ≥ 12 weeks.
4. Eastern Collaborative Oncology Group (ECOG) physical status score: 0 to 1.
5. B-cell non-Hodgkin's lymphoma expressing CD20 antigen clearly diagnosed by pathology
6. Patients with non-Hodgkin's lymphoma must have measurable lesions that meet the Lugano 2014 criteria for lymphoma efficacy assessment, requiring lymph node lesions >1.5 cm in either length or extra-nodal lesions >1.0 cm in either length.

Exclusion Criteria:

1. history of severe allergy or anaphylactic reaction to monoclonal antibody therapy (or recombinant antibody-associated fusion protein).
2. previous treatment with CD20-CD3 bispecific antibodies.
3. failure to resolve toxicity after prior antitumor therapy, i.e., no return to baseline or grade 0-1 as defined by NCI-CTCAE 5.0 (except for alopecia, hyperpigmentation). Irreversible toxicity that is not reasonably expected to be exacerbated by the study drug and may be enrolled upon confirmation with the sponsor.
4. Received antitumor therapy such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, or biologic therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose. Non-tumor related conditions that are amenable to hormone therapy (e.g. insulin therapy for diabetes and hormone replacement therapy).
5. receive autologous hematopoietic stem cell transplantation within 100 days prior to the first dose
6. have undergone, or are expected to require during the study period, major surgery (as judged by the investigator) or are recovering from surgery within 4 weeks prior to the first dose
7. active hepatitis B or C. Active hepatitis B defined as positive for hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) with HBV DNA above the upper limit of the study center's normal value; active hepatitis C defined as positive for hepatitis C antibody and HCV RNA above the upper limit of the study center's normal value.
8. history of cardiac disease: New York Heart Association (NYHA) > Class II congestive heart failure, myocardial infarction occurring within 6 months prior to enrollment, or arrhythmia requiring antiarrhythmic therapy and/or left ventricular ejection fraction < 50%.
9. two or more malignancies within 5 years prior to the first dose. Except for early malignancies that have been eradicated (carcinoma in situ or stage I tumors), such as adequately treated cervical carcinoma in situ, basal cell or squamous epithelial cell skin cancer.
10. persons with uncontrollable psychiatric disorders
11. patients with a history of drug abuse or alcohol abuse
12. other conditions judged by the investigator to be inappropriate for participation in this study, including but not limited to having any disease or medical history that may confound study results and interfere with patient compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
MTD | Throughout the dose escalation and dose expansion phases,, an average of 1.5 years
  It is suitable for dose escalation and dose extension.If the number of DLT patients is 0 and the next higher dose is unacceptable, the current dose is declared MTD.
RP2D | Throughout the dose escalation and dose expansion phases, an average of 1.5 years
  It is suitable for dose escalation and dose extension.RP2D will be determined based on a combination of safety, tolerability, PK and/or pharmacodynamic studies .

SECONDARY OUTCOMES:
DLT events | Up to 2 years
  Incidence and severity of DLT events.
Adverse events (AEs) | Up to 2 years
  Incidence and severity of adverse events (AEs)
Serious adverse events (SAEs) | Up to 2 years
  Incidence and severity of serious adverse events (SAEs).
abnormal changes in clinically significant laboratory tests and other examinations | Up to 2 years
  abnormal changes in clinically significant laboratory tests and other examinations
Objective Response Rate (ORR) | Up to 2 years
  Objective Response Rate (ORR) as Assessed by Investigator according to Lugano 2014
Complete Response (CR) | Up to 2 years
  Complete Response (CR) as Assessed by Investigator according to Lugano 2014
Duration of Objective Response (DOR) | Up to 2 years
  Duration of Objective Response (DOR) as Assessed by Investigator
Duration of Complete Response (DOCR) | Up to 2 years
  Duration of Complete Response (DOCR) as Assessed by Investigator
Time to Response(TTR) | Up to 2 years
  Time to Response(TTR) as Assessed by Investigator
Progression-Free Survival (PFS) | Up to 2 years
  Progression-Free Survival (PFS) as Determined by Investigator
Overall Survival (OS) | Up to 2 years
  Overall Survival (OS)
Antidrug antibodies (ADA) and/or neutralizing antibodies (Nab) | At pre-defined intervals up to 2 years
  incidence of antidrug antibodies (ADA) and/or neutralizing antibodies (Nab)
Total exposure(AUC) of JS203 | At pre-defined intervals up to 2 years
  Total exposure(AUC) of JS203
Maximum Plasma Concentration (Cmax) of JS203 | At pre-defined intervals up to 2 years
  Maximum Plasma Concentration (Cmax) of JS203
Half-life(T1/2) of JS203 | At pre-defined intervals up to 2 years
  Half-life(T1/2) of JS203
Clearance(CL) of JS203 | At pre-defined intervals up to 2 years
  Clearance(CL) of JS203
Volume of Distribution (Vss) of JS203 | At pre-defined intervals up to 2 years
  Volume of Distribution (Vss) of JS203
Pharmacodynamic (PD) characteristics | At pre-defined interval up to 2 years
  CD20 receptor occupancy rate in peripheral blood cells
Pharmacodynamic (PD) characteristics | At pre-defined interval up to 2 years
  Changes in peripheral blood immune cell subtypes (B cells, T cells) before and after drug administration.
Pharmacodynamic (PD) characteristics | At pre-defined interval up to 2 years
  Changes in peripheral blood cytokines (IL-2, IL-4, IL-6, IL-10, TNF-α, IFN-γ) before and after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China